CLINICAL TRIAL: NCT02967653
Title: Atorvastatin for the Treatment of Lithium-Induced Nephrogenic Diabetes Insipidus: A Randomized Controlled Trial
Brief Title: Atorvastatin for the Treatment of Lithium-Induced Nephrogenic Diabetes Insipidus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Dr. Karl Looper, Psychiatrist-in-Chief, Associate Professor, Dept. of Psychiatry, McGill University; Co-Lead, Geri-PARTy Research Group, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16/02
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Lithium Use, Nephrogenic Diabetes Insipidus
MeSH Terms: conditions — Diabetes Insipidus, Nephrogenic | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will be randomized to a placebo a day using simple 1:1 randomization using random.org, for 12 weeks.
  Interventions: Drug: Atorvastatin
- Atorvastatin (Experimental): Patients will be randomized to Atorvastatin 20mg/day for 12 weeks or pill placebo.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Member of drug class called statins, primarily used as a lipid-lowering agent and the prevention of events associated with cardiovascular disease
  Other Names: Lipitor

SUMMARY:
Lithium remains the gold-standard treatment for bipolar disorder, with 30-40% of patients with responding preferentially to this medication. Additionally, lithium is commonly used in treatment-resistant depression, and other psychiatric disorders (e.g. schizoaffective disorder). Lithium is especially valuable considering the great difficulty in achieving and maintaining symptomatic remission, the high rates of disability, as well as tremendous personal, family, and societal costs associated with bipolar disorder and treatment-resistant depression. Despite this, clinicians are increasingly avoiding lithium, largely due to fear of irreversible chronic kidney disease (CKD), particularly in North America.

It is well known that lithium exposure, even when dosed safely (<1.0mmol/L in adults 11 and <0.8mmol/L in geriatric patients 12,13), can increase the risk of CKD by 3 times, in large part through Nephrogenic Diabetes Insipidus (NDI) 14-19. NDI itself has also been associated with acute kidney injury 20, and life-threatening hypernatremia, which is an electrolyte imbalance characterized by high levels of blood sodium. Aside from hypertension, diabetes mellitus, aging, and other nonspecific CKD risk factors.

NDI is characterized by excessive thirst (polydipsia) due to increased production of dilute urine (polyuria). In NDI, lithium is believed to interact with the inositol monophosphate and protein kinase C pathways, thereby affecting calcium-related intracellular signaling, cyclic AMP (cAMP), inhibition of Glycogen Synthase Kinase-3 Beta (GSK3Beta), activation of MAP Kinase and many other pathways.

NDI occurs commonly in lithium users: 50% of chronic lithium users have urinary concentrating difficulties, with 12-19% have decreased urine osmolality (UOsm) <300mOsm/Kg).

To date, amiloride (5-20mg/day) is the only medication with prior evidence of therapeutic effectiveness in NDI from randomized clinical trials. However as a potassium-sparing diuretic 31, amiloride can lead to lithium-level elevations, and can thereby theoretically increase the risk of lithium-associated CNS and acute renal toxicity.

There is a need for novel, well-tolerated agents for the treatment of lithium-induced NDI.

We recently demonstrated that statins, which are well-tolerated and commonly used medications, are associated with low lithium-induced NDI risk in the first and only previous cross-sectional study examining statins and NDI in humans (n=71) 33. In this study we examined current lithium users aged 20-95, who had a mean lithium duration and serum lithium level of 10.6 years and 0.62mmol/L, respectively. Patients were assessed for UOsm following 10-hour water-restriction, a reliable measure of NDI. We found that 0% (0/17) of statin users compared to 20.4% (11/54) on non-users had UOsm <300mOsm/Kg following 10-hour water-restriction (Fisher's Exact p=0.055). The main statin prescribed in our previous study was atorvastatin 10-40mg/day (n=10) 33, which is the most widely used statin for cardiovascular disease. Atorvastatin and other statins are well-tolerated and have not been found to have adverse effects on mood, cognition, or renal function.

The mechanism by which statins may treat NDI is not yet known, but two independent mice studies have demonstrated the effectiveness of statins in treating genetic forms of NDI. In those mice models of genetic NDI, prostaglandin and intracellular cytoskeleton proteins pathways were thought to explain statins' activity on NDI.

In preparation for this project, our co-investigators Drs. Trepiccione and Christensen have initiated a pilot study in mice to investigate whether atorvastatin treatment could improve the lithium-induced NDI. NDI was induced in 10 mice by feeding mice with a LiCl-enriched diet for 15 days. After induction of NDI, a group of mice received intraperitoneal injection of atorvastatin (n=5) and a control group received vehicle (n=5) for additional 5 days in parallel with continued lithium treatment. Although our small statistical sample do not allow us to reach significance, (n=5 per group), the mice receiving atorvastatin showed a tendency to reduce polyuria.

In line with this research, our present research protocol aims at conducting a randomized controlled trial investigating a statin, such as atorvastatin, in the treatment of lithium-induced NDI.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 85 years of age
* Individuals with any psychiatric disorder who are taking lithium

  o Patients will be recruited from the Douglas Mental Health University Institute, Jewish General Hospital and McGill University Health Centre.
* Able and willing to give informed consent.
* Chronic and current lithium users (at least 2 months of Lithium use).
* Stable dose of lithium for the past 2 months.
* Patients taking any lithium level will be included.
* Patients with any psychiatric diagnosis will also be included.
* NDI defined as a 10-hour water restriction UOsm <600mOsm/Kg.

Exclusion Criteria:

* Patients allergic to Statins
* Patients with statin use within 6 weeks prior to the study
* Patients with a past history of severe adverse reaction to statins.
* Patients with a baseline Low Density Lipoprotein (LDL) level <1.5.
* Relative contraindications to statin use 42: pregnancy or lactation, concurrent use of fibrates, heavy ethanol consumption (>50 units/week).
* Incapacity to consent
* Deemed by the treating physician to have a severe cognitive or behavioural disturbance such as acute delirium or moderate-severe DSM5 Neurocognitive Disorder (dementia), preventing their ability to complete safely the study questionnaire and/or to provide blood and urine test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Raw Urine Osmolality value at 12 week follow-up, adjusted for baseline (UOsm in mOsm/Kg) | 12 weeks follow-up
  Urine Osmolality value at 12 week follow-up

SECONDARY OUTCOMES:
Raw aquaporins-2 (AQP-2) values at 12 week follow-up, adjusted for baseline | 12 weeks follow-up
  aquaporins-2 measurement as adjusted for baseline
Raw Urine Volume (mL/24h) value at 12 week follow-up, adjusted for baseline | 12 weeks follow-up
  24h urine volume values measured as adjusted for baseline
Raw Self-Reported Fluid Intake value 12 week follow-up, adjusted for baseline | 12 weeks follow-up
  self-reported fluid intake #measurement as adjusted for baseline

OTHER OUTCOMES:
Raw value of Cognition in the domain of executive function at 12 week follow-up, adjusted for baseline | 12 weeks follow-up
  Using Screen for Cognitive Impairment in Psychiatry (SCIP), Stroop, Trials A/Trials B tests
Safety Measures | 12 weeks follow-up
  Creatine kinase (CK) and Low Density Lipoprotein (LDL) Liver function tests Thyroid function (TSH) Calcium levels eGFR
Subgroup Analyses - Raw Urine Osmolality value at 12 week follow-up, adjusted for baseline in patients UOsm <300mOsm/Kg | 12 weeks follow-up
  Subgroup analyses

CONTACTS AND LOCATIONS:
Overall Officials: Soham F Rej, MD, M.Sc., Principal Investigator — Jewish General Hospital
Locations (3):
- Canada (3):
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fotso Soh J, Beaulieu S, Trepiccione F, Linnaranta O, Torres-Platas G, Platt RW, Renaud S, Su CL, Mucsi I, D'Apolito L, Mulsant BH, Levinson A, Saury S, Muller D, Schaffer A, Dols A, Low N, Cervantes P, Christensen BM, Herrmann N, Rajji T, Rej S. A double-blind, randomized, placebo-controlled pilot trial of atorvastatin for nephrogenic diabetes insipidus in lithium users. Bipolar Disord. 2021 Feb;23(1):66-75. doi: 10.1111/bdi.12973. Epub 2020 Jul 16. PMID 32621644
- [Derived] Fotso Soh J, Torres-Platas SG, Beaulieu S, Mantere O, Platt R, Mucsi I, Saury S, Renaud S, Levinson A, Andreazza AC, Mulsant BH, Muller D, Schaffer A, Dols A, Cervantes P, Low NC, Herrmann N, Christensen BM, Trepiccione F, Rajji T, Rej S. Atorvastatin in the treatment of Lithium-induced nephrogenic diabetes insipidus: the protocol of a randomized controlled trial. BMC Psychiatry. 2018 Jul 16;18(1):227. doi: 10.1186/s12888-018-1793-9. PMID 30012135